CLINICAL TRIAL: NCT05107960
Title: Special Drug Use Surveillance; AZILVA Tablets and AZILVA Granules 1% in Pediatric Use
Brief Title: A Study of Azilsartan in Children From 6 to Less Than 16 Years Old With High Blood Pressure
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-536-4001; jRCT2031210414 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-10-28; First posted 2021-11-04 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — azilsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Azilsartan: Azilsartan tablets or granules formulation, orally once daily. For children aged 6 years or older, the usual initial oral dosage of azilsartan is 2.5 mg and 5 mg once daily for those weighing <50 kg and >=50 kg, respectively.
  Interventions: Drug: Azilsartan (TAK-536)

INTERVENTIONS:
Drug: Azilsartan (TAK-536) — Azilsartan Tablets, Azilsartan Granules
  Other Names: AZILVA Tablets, AZILVA Granules 1%

SUMMARY:
The main aim of this study is to check for side effects from treatment with azilsartan and how well azilsartan controls blood pressure in children from 6 to less than 16 years old with high blood pressure.

The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

During the study, participants with high blood pressure will take azilsartan tablets or azilsartan granules once a day according to their clinic's standard practice. The study doctors will check for side effects from azilsartan for up to 12 months after treatment starts.

ELIGIBILITY:
Inclusion Criteria

1. Participants aged 6 years or older and less than 16 years
2. Participants with hypertension

Exclusion Criteria Participants with contraindications to azilsartan.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with hypertension aged 6 years or older and less than 16 years will be included in the survey.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites).

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/618bf1c5f571d4002a64b390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the survey at 3 investigative sites in Japan, from 16 December 2021 to 24 August 2024.
Pre-assignment Details: Participants with high blood pressure who received azilsartan tablets or granules formulation were enrolled. Participants received azilsartan as part of a routine medical care.
Groups:
- Azilsartan: Participants received azilsartan tablets or granules formulation orally, once daily as part of routine medical care. For children aged 6 years or older, the usual initial oral dosage of azilsartan was 2.5 mg once daily for those weighing <50 kg and 5 mg once daily for those weighing >=50 kg, respectively.
Period: Overall Study
Arm/Group | Azilsartan
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (1.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product. It does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product (including an investigational product for a new indication in Japan), whether or not related to the pharmaceutical product. For regenerative medicine products, any failure report is also handled as an adverse event.
Time Frame: Up to Months 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
Participants | 0

2. Primary Outcome: Number of Participants Who Experienced at Least One Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability /incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Up to Months 12
Population: Safety Analysis Set, The safety analysis set was defined as all participants who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Mean Value of Systolic Blood Pressure
Time Frame: Up to 12 Months
Population: Efficacy analysis set: The efficacy analysis set was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. The analyzed numbers were participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
mmHg
  Baseline | 121.8 (10.47)
  Month 1: number analyzed (Participants) | 4
  Month 1 | 109.8 (17.90)
  Month 2: number analyzed (Participants) | 3
  Month 2 | 112.3 (24.01)
  Month 3: number analyzed (Participants) | 2
  Month 3 | 117.5 (20.51)
  Month 4: number analyzed (Participants) | 4
  Month 4 | 113.3 (6.90)
  Month 5: number analyzed (Participants) | 2
  Month 5 | 115.5 (3.54)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 97.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 7: number analyzed (Participants) | 2
  Month 7 | 116.5 (13.44)
  Month 8: number analyzed (Participants) | 1
  Month 8 | 116.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 9: number analyzed (Participants) | 1
  Month 9 | 102.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 10: number analyzed (Participants) | 0
  Month 11: number analyzed (Participants) | 2
  Month 11 | 108.5 (12.02)
  Month 12: number analyzed (Participants) | 0

4. Primary Outcome: Mean Value of Diastolic Blood Pressure
Time Frame: Up to 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
mmHg
  Baseline | 72.8 (10.31)
  Month 1: number analyzed (Participants) | 4
  Month 1 | 65.8 (9.78)
  Month 2: number analyzed (Participants) | 3
  Month 2 | 68.0 (12.00)
  Month 3: number analyzed (Participants) | 2
  Month 3 | 77.5 (3.54)
  Month 4: number analyzed (Participants) | 4
  Month 4 | 64.0 (8.76)
  Month 5: number analyzed (Participants) | 2
  Month 5 | 58.5 (0.71)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 61.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 7: number analyzed (Participants) | 2
  Month 7 | 57.0 (11.31)
  Month 8: number analyzed (Participants) | 1
  Month 8 | 66.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 9: number analyzed (Participants) | 1
  Month 9 | 51.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 10: number analyzed (Participants) | 0
  Month 11: number analyzed (Participants) | 2
  Month 11 | 57.0 (0.00)
  Month 12: number analyzed (Participants) | 0

5. Primary Outcome: Change From Baseline in Mean Value of Systolic Blood Pressure
Time Frame: Baseline, Up to 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
mmHg
  Month 1: number analyzed (Participants) | 4
  Month 1 | -8.5 (24.80)
  Month 2: number analyzed (Participants) | 3
  Month 2 | -14.7 (30.01)
  Month 3: number analyzed (Participants) | 2
  Month 3 | 2.5 (20.51)
  Month 4: number analyzed (Participants) | 4
  Month 4 | -5.0 (14.45)
  Month 5: number analyzed (Participants) | 2
  Month 5 | -10.0 (11.31)
  Month 6: number analyzed (Participants) | 1
  Month 6 | -33.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 7: number analyzed (Participants) | 2
  Month 7 | -9.0 (1.41)
  Month 8: number analyzed (Participants) | 1
  Month 8 | -14.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 9: number analyzed (Participants) | 1
  Month 9 | -34.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 10: number analyzed (Participants) | 0
  Month 11: number analyzed (Participants) | 1
  Month 11 | -24.5 (7.78)
  Month 12: number analyzed (Participants) | 0

6. Primary Outcome: Change From Baseline in Mean Value of Diastolic Blood Pressure
Time Frame: Baseline, Up to 12 Months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan
Number analyzed (Participants) | 5
mmHg
  Month 1: number analyzed (Participants) | 4
  Month 1 | -9.0 (14.90)
  Month 2: number analyzed (Participants) | 3
  Month 2 | -3.3 (23.16)
  Month 3: number analyzed (Participants) | 2
  Month 3 | 12.0 (1.41)
  Month 4: number analyzed (Participants) | 4
  Month 4 | -10.8 (13.89)
  Month 5: number analyzed (Participants) | 2
  Month 5 | -6.0 (1.41)
  Month 6: number analyzed (Participants) | 1
  Month 6 | -24.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 7: number analyzed (Participants) | 2
  Month 7 | -7.5 (10.61)
  Month 8: number analyzed (Participants) | 1
  Month 8 | -19.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 9: number analyzed (Participants) | 1
  Month 9 | -14.0 (NA) — The standard deviation was not evaluable due to low number of participants with events.
  Month 10: number analyzed (Participants) | 0
  Month 11: number analyzed (Participants) | 2
  Month 11 | -18.0 (14.14)
  Month 12: number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 12 Months
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to the survey treatment.
Arm/Group | Azilsartan
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT05107960/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT05107960/SAP_001.pdf